CLINICAL TRIAL: NCT06490627
Title: Unraveling the Impact of Thalidomide at Diverse Doses in Transfusion Dependent Beta Thalassemia
Acronym: BTM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Responsible Party: Principal Investigator, Safia mehmood khan, Doctor, National Institute of Blood Disease Center, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBD/IRB-266/01-2024
Record Dates: First submitted 2024-06-20; First posted 2024-07-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Fetal Hemoglobin; Thalassemia Major; Genetic Disease
Keywords: thalidomide; safety and efficacy; thalassemia; fetal hemoglobin inducer
MeSH Terms: conditions — beta-Thalassemia; Genetic Diseases, Inborn; Thalassemia | interventions — Thalidomide

STUDY DESIGN:
Intervention Model Description: in this study three groups have been made. one is control group which received no intervention and on transfusion only. whereas other two groups are interventional both received thalidomide. one received thalidomide at 5-6mg/kg/day and second at 7-8 mg/kg/day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): in this group, patient will not receive any interventional drug or treatment drug so simply they will blood transfusion dependent.
- Group 1 Thalidomide (Experimental): In this group , thalassemia patients will receive thalidomide at the dose of 5-6mg/kg/day at night with aspirin.
  Interventions: Drug: Thalidomide
- Group 2 Thalidomide (Active Comparator): In this group , thalassemia patients will receive thalidomide at the dose of 7-8mg/kg/day at night with aspirin
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Thalidomide is being investigated for its therapeutic efficacy and safety profile in transfusion-dependent beta thalassemia patients.
  Participants in this arm received thalidomide. Thalidomide was administered orally at a dosage of 5-6mg/kg/day. The medication was taken continuously or on a specified schedule (e.g., daily,) for the duration of the study period, which lasted 2 years. Participants were monitored for adherence to the medication regimen and for any adverse effects throughout the intervention period.
  Arms: Group 1 Thalidomide
Drug: Thalidomide — Thalidomide is being investigated for its therapeutic efficacy and safety profile in transfusion-dependent beta thalassemia patients.
  Participants in this arm received thalidomide. Thalidomide was administered orally at a dosage of 7-8mg/kg/day. The medication was taken continuously or on a specified schedule (e.g., daily,) for the duration of the study period, which lasted 2 years. Participants were monitored for adherence to the medication regimen and for any adverse effects throughout the intervention period.
  Arms: Group 2 Thalidomide

SUMMARY:
The project "Unraveling the Impact of Thalidomide at Diverse Doses in Transfusion Dependent Beta Thalassemia" investigates the safety and efficacy of low-dose thalidomide in managing beta thalassemia, a genetic disorder causing anemia. Conducted over two years at NIBD hospital, the study involves 54 transfusion-dependent patients aged 8-35. The primary objective is to correlate thalidomide doses with disease severity, adverse effects, and treatment response, aiming to optimize treatment strategies and reduce side effects.

Data will be collected through clinical interviews and medical record reviews and analyzed using SPSS. Key variables include hemoglobin levels, leukocyte and reticulocyte counts, platelets, liver and spleen size, genetic modifiers, and transfusion frequency. Inclusion criteria are specific to beta thalassemia patients, while exclusion criteria rule out those with liver dysfunction, married patients, lactating mothers, and those with a history of thrombosis or fits.

DETAILED DESCRIPTION:
Thalassemia is an inherited monogenic blood disorder caused by improper synthesis of the hemoglobin chain, inherited in an autosomal recessive pattern. Hemoglobin is essential for oxygen transport from the lungs to body tissues. Initially observed in individuals of Italian descent, thalassemia is characterized by anemia, enlarged spleen, and bone abnormalities. It affects approximately 1.5% of the global population, with 60,000 infants born annually with severe forms such as homozygous alpha thalassemia, beta-thalassemia, and HbH disease. Patients with thalassemia major require frequent blood transfusions and iron chelation therapy to manage iron overload, which can lead to complications like cirrhosis, heart failure, and growth retardation. Iron chelators such as deferasirox, deferiprone, and deferoxamine are used in Pakistan either as solo or combination therapy based on iron levels. Bone marrow transplantation from HLA-identical siblings offers a curative option with high success rates, but non-HLA identical cases are less promising. Emerging therapies like HbF production reactivation, cell therapy, and gene therapy show potential for better management of thalassemia.

Beta thalassemia is a prevalent genetic disorder, especially in the Mediterranean, Middle East, and Southeast Asia. It causes reduced hemoglobin production, severe anemia, and dependence on regular blood transfusions, which lead to iron overload and associated complications. Thalidomide, initially marketed as a sedative in 1954 and later withdrawn due to teratogenic effects, has shown efficacy in hematologic disorders. Its potential in beta thalassemia, particularly for reducing transfusion requirements and managing iron overload, remains underexplored. Preliminary studies suggest thalidomide could reduce transfusion needs, but comprehensive dose-dependent research is lacking. This study aims to evaluate the effects of thalidomide at various doses in transfusion-dependent beta thalassemia patients, hypothesizing that optimal dosing can improve disease management and quality of life.

Preliminary research indicates thalidomide might reduce transfusion frequency and manage iron overload in beta thalassemia patients. However, detailed dose-dependent studies are necessary. This research aims to fill the gap by exploring thalidomide's benefits and safety profiles at diverse doses, potentially revolutionizing the therapeutic approach to beta thalassemia.

The study aims to evaluate the impact of diverse thalidomide doses on reducing transfusion dependency in beta thalassemia patients. Primary objectives include assessing the efficacy of thalidomide in reducing transfusion needs. Secondary objectives involve evaluating the impact on complete blood count, liver function, spleen size, serum ferritin levels, and iron overload, alongside monitoring safety profiles and adverse events. Impact of genetic modifiers on thalidomide and beta thalassemia phenotype will also monitor in this study.

The study will be a single-center randomized controlled clinical trial at the National Institute of Blood Disease and Bone Marrow Transplant Hospital in Karachi, Pakistan, specializing in genetic disorders and hematology-oncology. Participants will be divided into treatment (with two dose groups) and control groups, with a total sample size of 54 calculated using OpenEpi. The study will span two years, from May 2024 to May 2026, involving data collection through medical records, interviews, and questionnaires. Ethical approval and informed consent will be obtained, ensuring patient confidentiality and adherence to ethical standards.

Data will include patient demographics (age, gender, ethnicity, marital status, weight, height), clinical variables (type of thalassemia, comorbidities, previous treatment), laboratory variables (hemoglobin, leukocyte count, reticulocyte count, platelets, lactate dehydrogenase, ferritin, d-dimer, bilirubin levels, SGPT), genetic modifiers (HBB mutation, XMN polymorphism, BCL11A polymorphism, alpha chain co-inheritance), and others (spleen and liver size, fibroscan, T2 star, transfusion frequency).

ELIGIBILITY:
Inclusion Criteria:

* Know case of beta thalassemia major/ intermediate ( transfusion dependent)
* willing to give informed consent

Exclusion Criteria:

* Patients with comorbidities such as liver dysfunction
* Married patients
* Lactating mother
* H/O thrombosis and fits

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
transfusion dependency | 1 year
  Transfusion frequency will be assessed by recording the number of blood transfusions a patient receives over a specified period, such as weekly, monthly, or annually. This data will be collected from patient medical records and/or transfusion logs, ensuring accurate tracking of each transfusion event

SECONDARY OUTCOMES:
hemoglobin levels. | 2 years
  Hemoglobin levels will be assessed using a complete blood count (CBC) test, measured in grams per deciliter (g/dL) of blood. This test is conducted through a venous blood sample, which is then analyzed using an automated hematology analyzer to determine the hemoglobin concentration.
total leukocyte count. | 2 years
  Leukocyte count will be assessed using a complete blood count (CBC) test, measured in thousands of cells per microliter (thousand cells/µL) of blood. This test involves analyzing a venous blood sample with an automated hematology analyzer to determine the total number of white blood cells present.
reticulocyte count | 2 years
  Reticulocyte count will be assessed using a complete blood count (CBC) test, measured as a percentage of the total red blood cells or as an absolute number per microliter (µL) of blood. This test involves analyzing a venous blood sample with an automated hematology analyzer, which identifies and quantifies reticulocytes using specific staining techniques.
Platelets | 2 years
  Platelet count will be assessed using a complete blood count (CBC) test, measured in thousands of cells per microliter (thousand cells/µL) of blood. This test involves analyzing a venous blood sample with an automated hematology analyzer to determine the number of platelets.
impact of genetic modifiers (e.g., HBB mutation, XMN polymorphism, BCL11A polymorphism, and co-inheritance of alpha chain) on the treatment outcomes with thalidomide. | 2 years
  Genetic modifiers will be assessed through genetic testing E.g thalassemia genetic profile, focusing on specific genes or genetic variations known to influence the expression or function of proteins related to the condition under study. This analysis helps identify how genetic factors may modify disease progression, treatment response, or other relevant outcomes.
Spleen Size | 2 years
  Spleen size will be assessed using imaging techniques such as ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI). Measurements will be reported in centimeters (cm).
Serum Glutamate Pyruvate Transaminase, | 2 years
  Serum Glutamate Pyruvate Transaminase, also known as alanine aminotransferase (ALT), will be assessed through a blood test, measured in units per liter (U/L). This test analyzes a venous blood sample to determine the concentration of ALT, an enzyme primarily found in the liver cells.
Serum Ferritin Levels | 2 years
  Serum ferritin levels will be assessed using a blood test, measured in nanograms per milliliter (ng/mL). A venous blood sample will be analyzed in a clinical laboratory using immunoassay techniques to determine the concentration of ferritin, providing an indicator of the body's iron stores.
lactate dehydrogenase | 2 years
  Lactate dehydrogenase (LDH) levels will be assessed through a blood test, measured in units per liter (U/L). This test analyzes a venous blood sample to determine the concentration of LDH, an enzyme involved in cellular metabolism. Elevated LDH levels may indicate tissue damage or disease,
Nucleated red blood cells | 2 years
  Nucleated red blood cells (NRBCs) will be assessed using a complete blood count (CBC) test with a differential, measured as the number of NRBCs per 100 white blood cells (WBCs) or as an absolute number per microliter (µL) of blood. This test involves analyzing a venous blood sample with an automated hematology analyzer, which can differentiate and count NRBCs to provide insights into bone marrow function and potential hematologic disorders.
D-dimer | 2 years
  D-dimer levels will be assessed through a blood test, typically measured in nanograms per milliliter (ng/mL) or micrograms per liter (µg/L). This test analyzes a venous blood sample to determine the concentration of D-dimer, a fibrin degradation product.
Total bilirubin | 2 years
  Total bilirubin (TBIL) levels will be assessed through a blood test, measured in milligrams per deciliter (mg/dL). This test analyzes a venous blood sample to determine the total concentration of bilirubin, including both direct (conjugated) and indirect (unconjugated) bilirubin.
Indirect bilirubin | 2 years
  Indirect bilirubin (IBIL) levels will be assessed through a blood test, measured in milligrams per deciliter (mg/dL). This test analyzes a venous blood sample to determine the concentration of unconjugated bilirubin, which is a byproduct of red blood cell breakdown before it is processed by the liver.
Fibroscan | 2 years
  FibroScan will be used to assess liver stiffness and steatosis, which can be indicative of liver iron overload. Elevated serum ferritin levels may suggest iron accumulation in the liver, and FibroScan provides a non-invasive method to evaluate the extent of liver fibrosis and fat content.
T2 star imaging | 2 years
  T2* (T2 star) magnetic resonance imaging (MRI) will be used to assess liver iron concentration in relation to serum ferritin levels. This imaging technique measures the rate of signal decay in liver tissue, which is inversely correlated with iron content. A shorter T2* value indicates higher iron concentration. T2* MRI provides a non-invasive, quantitative assessment of liver iron overload.
transfusion dependency | 2 year
  Transfusion frequency will be assessed by recording the number of blood transfusions a patient receives over a specified period, such as weekly, monthly, or annually. This data will be collected from patient medical records and/or transfusion logs, ensuring accurate tracking of each transfusion event

OTHER OUTCOMES:
Safety Profile: | 2 years
  The safety profile will be assessed by monitoring and documenting adverse events, side effects, and any other safety-related outcomes throughout the study period. This includes recording and analyzing data on patient-reported symptoms, clinical observations, laboratory test results (including those for the parameters previously discussed like liver enzymes, kidney function tests, etc.), and any other relevant safety assessments specified in the study protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of blood disease and bone marrow transplant, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Maybe i will share the IPD upon request

REFERENCES:
- [Background] Swabb EA, Sugerman AA, Platt TB, Pilkiewicz FG, Frantz M. Single-dose pharmacokinetics of the monobactam azthreonam (SQ 26,776) in healthy subjects. Antimicrob Agents Chemother. 1982 Jun;21(6):944-9. doi: 10.1128/AAC.21.6.944. PMID 7202343